CLINICAL TRIAL: NCT00895830
Title: Randomised, Double-blind, Placebo-controlled, Phase II Study to Assess the Safety and Efficacy of Different Doses of Intravenous APD405 for the Prevention of Post-operative Nausea and Vomiting
Brief Title: Dose-ranging Study of APD405 in Post-operative Nausea and Vomiting (PONV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Chief Medical Officer, Acacia Pharma Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DP10002
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental): 0.3mg dose level
  Interventions: Drug: APD405
- 3 (Experimental): 1mg dose level
  Interventions: Drug: APD405
- 4 (Experimental): 2mg dose level
  Interventions: Drug: APD405
- 5 (Experimental): 3mg dose level
  Interventions: Drug: APD405

INTERVENTIONS:
Drug: APD405 — IV
  Arms: 2; 3; 4; 5
Drug: Placebo — IV
  Arms: 1

SUMMARY:
To assess the efficacy and safety of different doses of APD405 in the prevention of post-operative nausea and vomiting (PONV) in adult patients at moderate to high-risk of PONV. Patients must be undergoing elective surgery under general anaesthesia (hysterectomy (any surgical technique), cholecystectomy (any surgical technique) or "other" elective surgery scheduled to last at least one hour from induction of anaesthesia), requiring at least one overnight stay in hospital, and have at least 2 of the following risk factors for PONV: Past history of PONV and/or motion sickness; Non-smoking status; Female gender; Planned opiate use for post-operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Written informed consent
* Patients undergoing elective surgery under general anaesthesia requiring at least one overnight stay in hospital for either:

  1. Hysterectomy (any surgical technique)
  2. Cholecystectomy (any surgical technique)
  3. Other elective surgery requiring overnight admission to hospital and scheduled to last at least 1 hour from induction of anaesthesia
* Patients with at least 2 risk factors for PONV, defined as 2 of the following:

  1. Past history of PONV and/or motion sickness
  2. Non-smoking status
  3. Female gender
  4. Planned opiate use for post-operative analgesia
* American Society of Anesthesiologists (ASA) risk score I-III (see Appendix 3)
* Adequate hepatic and renal function

  * Alanine aminotransferase (ALT) <2.5 * upper limit normal (ULN)
  * Aspartate aminotransferase (AST) <2.5 * ULN
  * Bilirubin <1.5 * ULN
  * Creatinine <1.5 * ULN
* Adequate haematological function

  * Haemoglobin ≥9.5 g/dL
  * White blood count 4.0-11.0 * 10^9/L
  * Platelet count ≥150 - 400 * 10^9/L
* Ability and willingness to give written informed consent

Exclusion Criteria:

* Patients undergoing outpatient/day case surgery
* Patients undergoing surgery where the patient is expected to remain ventilated for a period after surgery
* Patients undergoing intra-thoracic, transplant or central nervous system surgery
* Patients receiving a local anaesthetic/regional neuraxial (intrathecal or epidural) block
* Patients receiving monoamine oxidase inhibitor (MAOI) therapy currently or in the preceding 3 weeks
* Patients with a pre-existing vestibular disorder or history of dizziness
* Patients that are expected to need a naso- or oral-gastric tube in situ after surgery is completed
* Any other concurrent disease or illness that, in the opinion of the investigator makes the patient unsuitable for the study
* Patients treated with regular anti-emetic therapy including corticosteroids
* Patients receiving CYP3A4 inducers or inhibitors within 7 days prior to study including but not limited to erythromycin, itraconazole, nefazodone, diltiazem, verapamil, rifampicin
* Patients with pre-existing nausea or vomiting 24 hours before surgery
* Patients who are breast feeding or pregnant
* Patients with a history of alcohol abuse
* Patients diagnosed with Parkinson's disease
* Patients who have received anti-cancer chemotherapy in the previous 4 weeks
* Patients with pre-existing clinically significant cardiac arrhythmia
* Patients with a history of epilepsy
* Patients who have participated in a previous study within the last 28 days (French sites only: Patients who have participated in a previous study within the last 6 months, if required by national or local regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tramèr, MD, Principal Investigator — University Hospital, Geneva
Locations (18):
- United States (3):
  - UCSF Medical Center at Mt Zion, San Francisco, California
  - Duke University Medical Center, Durham, North Carolina
  - Memorial Hermann-Memorial City Hospital, Houston, Texas
- France (7):
  - University Hospital, Besançon
  - Hôpital mère enfant, Bron
  - Hôpital Huriez, Lille
  - University Hospital, Nancy
  - Hôpital FOCH, Paris
  - University Hospital, Reims
  - Hautepierre Hospital, Strasbourg
- Germany (6):
  - Charité - Universitätsmedizin, Berlin
  - Universität Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
  - Klinikum Ludwigshafen, Ludwigshafen
  - Philipps University, Marburg
  - University Hospitals of Würzburg, Würzburg
- Switzerland (2):
  - Geneva University Hospitals, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Derived] Kranke P, Rohm KD, Diemunsch P, Gan TJ, Apfel CC, Eberhart L, Minkowitz HS, Wallenborn J, Chassard D, Lebuffe G, Fox GM, Tramer MR. Intravenous buspirone for the prevention of postoperative nausea and vomiting. Eur J Clin Pharmacol. 2012 Nov;68(11):1465-72. doi: 10.1007/s00228-012-1284-8. Epub 2012 May 1. PMID 22546895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | APD405 0.3mg Dose | APD405 1mg Dose | APD405 2mg Dose | APD405 3mg Dose
Started | 51 | 50 | 49 | 52 | 55
Completed | 51 | 50 | 49 | 52 | 55
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | APD405 0.3mg Dose | APD405 1mg Dose | APD405 2mg Dose | APD405 3mg Dose | Total
Number analyzed (Participants) | 51 | 50 | 49 | 52 | 55 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.828) | 49.4 (13.575) | 49.5 (13.949) | 52.3 (16.191) | 50.3 (13.599) | 50.55 (14.198)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 49 | 43 | 45 | 49 | 231
  Male | 6 | 1 | 6 | 7 | 6 | 26
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 9 | 6 | 9 | 39
  France | 16 | 15 | 14 | 16 | 16 | 77
  Germany | 26 | 28 | 26 | 29 | 29 | 138
  Switzerland | 1 | 0 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Experienced Post-operative Nausea or Vomiting
Time Frame: 24 hours
Population: ITT
Measure: Number; unit: participants
Arm/Group | Placebo | APD405 0.3mg Dose | APD405 1mg Dose | APD405 2mg Dose | APD405 3mg Dose
Number analyzed (Participants) | 51 | 50 | 49 | 52 | 55
participants | 25 | 29 | 20 | 30 | 28

ADVERSE EVENTS:
Arm/Group | Placebo | APD405 0.3mg Dose | APD405 1mg Dose | APD405 2mg Dose | APD405 3mg Dose
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/50 | 2/49 | 2/52 | 3/55
Other Adverse Events (participants affected / at risk) | 46/51 | 46/50 | 45/49 | 45/52 | 51/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | APD405 0.3mg Dose (N=50) | APD405 1mg Dose (N=49) | APD405 2mg Dose (N=52) | APD405 3mg Dose (N=55)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-operative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | APD405 0.3mg Dose (N=50) | APD405 1mg Dose (N=49) | APD405 2mg Dose (N=52) | APD405 3mg Dose (N=55)
Procedural pain (Injury, poisoning and procedural complications) | 24 | 25 | 32 | 25 | 24
Nausea (Gastrointestinal disorders) | 26 | 28 | 20 | 30 | 25
Vomiting (Gastrointestinal disorders) | 15 | 13 | 13 | 22 | 18
Flatulence (Gastrointestinal disorders) | 5 | 7 | 7 | 7 | 4
Insomnia (Psychiatric disorders) | 6 | 3 | 8 | 7 | 6
Constipation (Gastrointestinal disorders) | 4 | 5 | 5 | 4 | 5
Hypertension (Vascular disorders) | 2 | 0 | 1 | 4 | 4
Hyp0kalaemia (Investigations) | 3 | 1 | 3 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 4 | 4 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No